CLINICAL TRIAL: NCT05827432
Title: Field-Cycling Imaging Effectiveness in Non-alcoholic Fatty Liver Disease Stratification
Brief Title: FCI Effectiveness in NAFLD Stratification
Acronym: FIELDS
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study suspended until new FCI scanner is operational.
Sponsor: NHS Grampian (Other Government)
Collaborators: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1-100-22
Record Dates: First submitted 2023-03-10; First posted 2023-04-25 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: Non-Alcoholic Fatty Liver Disease; Field-cycling imaging
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NAFLD (Experimental): Participants with different degree of steatohepatitis and NAFLD will undergo one FCI scan.
  Interventions: Device: Field-cycling imaging (FCI)

INTERVENTIONS:
Device: Field-cycling imaging (FCI) — FCI scan

SUMMARY:
The goal of this pilot study is exploring whether field-cycling imaging may be able to detect characteristics of liver disease in patients with different degree of non-alcoholic fatty liver disease (NAFLD) that could be important in reflecting disease progression.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) encompasses a spectrum of diseases extending from simple steatosis to non-alcoholic steatohepatitis (NASH), fibrosis, cirrhosis, and hepatocellular carcinoma (HCC). Currently, there is a pressing unmet clinical need to develop an effective non-invasive method to differentiate between different types of NAFLD and to support the initiation and monitoring of treatments designed to slow or halt progression of the disease.

Field-cycling imaging (FCI) is an innovative imaging technology pioneered at the University of Aberdeen. It has the ability to image human tissues non-invasively over a wide range of magnetic field strengths, directly informing on multi-scale tissue structure from nanometres to micrometres. This is not possible with traditional MRI. The potential of FCI in imaging NAFLD is particularly promising, due to its high sensitivity in quantifying and distinguishing protein content from fat.

The purpose of this pilot study is exploring whether FCI may be able to detect characteristics of liver disease, in patients with different degree of steatohepatitis and NAFLD, that could be important in reflecting progression of steatosis to liver fibrosis and HCC thereby potentially offering new diagnostic information that cannot be readily obtained with currently available imaging techniques.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a diagnosis of NAFLD
* Participants must be aged 18 and above
* Participants who meet the safety criteria for undergoing an MRI scan
* Participants who are able to fit inside the scanner
* Participants must be able to give fully informed consent
* Participants must be mobile enough to be positioned onto the FCI scanner couch

Exclusion Criteria:

* MRI-incompatible conditions, as detected in the MRI safety screening sheet
* Participants under 18 years old
* Participants who are unable to communicate in English
* Participants who are unable to give fully informed consent
* Women who are pregnant
* Restrictions to mobility that would prevent the correct positioning in the scanner
* Participants who suffer from claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Differentiation of NAFLD types, from steatosis to liver fibrosis, assessed by Field-Cycling Imaging (FCI) scan | At baseline
  Validation of FCI T1 dispersion profiles as a non-invasive technology to map out structural information on NAFLD that is not available by standard methods, by distinguishing protein content from fat, with application for medical research.

SECONDARY OUTCOMES:
NAFLD progression assessed by Field-Cycling Imaging (FCI) T1 dispersion profiles of liver tissue | At baseline
  Exploring the effectiveness of FCI T1 dispersion profiles of liver protein content, fat content, and fibrotic tissue in participants with NAFLD as a method for non-invasive assessment of disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Ashis Mukhopadhya, Dr, Principal Investigator — NHS Grampian
Locations (1):
- Aberdeen Royal Infirmary, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No